CLINICAL TRIAL: NCT01705171
Title: Is the Expression of the GLUT5 Specific Fructose Transport Protein Abnormal in Patients With Fructose Intolerance?
Status: Completed | Type: Observational
Sponsor: Brain-Gut Research Group (Other)
Responsible Party: Principal Investigator, C. Wilder-Smith, Dr. med., Brain-Gut Research Group
Other Study IDs: GGP1345012; GLUT5 (Other: Brain-Gut Research Group)
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Irritable Bowel Syndrome; Fructose Intolerance
Keywords: IBS; fructose intolerance; GLUT 5; GLUT 2
MeSH Terms: conditions — Irritable Bowel Syndrome; Fructose Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IBS patients with fructose intolerance: analysis of biopsies
- Control group: no IBS or fructose intolerance: analysis of biopsies

SUMMARY:
In this study we will investigate the expression of the fructose transport protein GLUT5 in the small intestine in patients with functional GI disoders and fructose intolerance compared to matched healthy controls.

DETAILED DESCRIPTION:
Intolerances to food are a major complaint of patients with functional gastrointestinal disorders (FGID) and even commoner in patients with inflammatory bowel disorders (IBD) (Barrett JS et al. Aliment Pharmacol Therap 2009;30:165-174). The most common forms of food intolerance are FODMAP (fermentable oligo-, di- and monosaccharide and polyol) -related, of which fructose and lactose are the best known. The prevalence of lactose and fructose intolerance in IBS patients is between 50 and 70% (Wilder-Smith CH et al. Gastroenterology 2009;136 (Suppl. 1): A324). Recent high quality studies have shown that the reduction of ingested FODMAP can lead to significant and long-term symptom improvement in patients shown to be intolerant by breath-testing. While the pathophysiology behind lactose intolerance is the reduction in small intestinal lactase availability, the mechanism in fructose intolerance and its relationship to malabsorption are unknown. One possible and so far uninvestigated mechanism is a reduction in the expression or activity of the specific fructose transporter, GLUT5, which is mainly responsible for luminal absorption of fructose. GLUT5 is mainly found in the small intestine, as well as various extra-intestinal organs. The clinical relevance of GLUT5 expression for food intolerances in humans has not been reported, but in a mouse model deletion of GLUT5 led to decreased absorption of dietary fructose and typical signs of malabsorption (Barone S et al. J Biol Chem 2009;284:5056-5066). The control of GLUT5 is dynamic and considerable upregulation together with increased absorption of fructose is evident in diabetes mellitus, while expression is decreased by inflammation and lipopolysaccharide endotoxin, an integral component of the outer membrane of all gram-negative bacteria, through the action of pro-inflammatory cytokines, such as TFN-a.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our practice for evaluation of symptoms consistent with FGID undergoing upper GI endoscopy with biopsy and fructose breath testing as part of their usual clinical evaluation. Male or female patients aged between 18 and 60 years with FGID (Irritable Bowel Syndrome (IBS), Functional Dyspepsia (FD) or Functional Bloating (FB), as defined by Rome III criteria.
* Successive patients without fructose intolerance undergoing upper GI endoscopy for other reasons without inflammatory disease

Exclusion Criteria:

* Inflammatory GI disease, coeliac's disease, other relevant systemic disorders as judged by investigator, concomitant antiinflammtory treatments, absent informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients referred to our practice for evaluation of symptoms consistent with FGID undergoing upper GI endoscopy with biopsy and fructose breath testing as part of their usual clinical evaluation.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
mRNA and protein expression of Glut5 | on day of endoscopy

SECONDARY OUTCOMES:
mRNA and protein expression of Glut2 | on day of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: C Wilder-Smith, MD, Principal Investigator — Brain-Gut Research Group
Locations (1):
- Gastoenterology Group Practice, Bern, Switzerland